CLINICAL TRIAL: NCT02656940
Title: Effects of Dietary Lipid Modulation in Energy Expenditure, Body Composition, Obesity-related Biomarkers and Gene Expression of Peroxisome Proliferator-Activated Receptors Alpha and Gamma 2 in Adipose Tissue of Obese Women
Brief Title: Dietary Lipids, Energy Expenditure and Obesity Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Vanessa Chaia Kaippert, Doctor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 778/10 Parecer CEP
Record Dates: First submitted 2016-01-07; First posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: obesity; lipids; energy expenditure; gene expression
MeSH Terms: conditions — Obesity | interventions — Fatty Acids, Monounsaturated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 - diet rich in n-3 and n-6 PUFA (Experimental): Assigned intervention: The dietary intervention was conducted by 60 days. Were prescribed normocaloric diets with similar macronutrient composition, varying only the type of lipids offered.
  Group 1 received diet rich in n-3 and n-6 polyunsaturated fatty acids (PUFA). The volunteers were asked to consume daily a mixture of virgin olive oil and soybean oil, totaling 35.2g to 52.8g, and 2 g of fish oil.
  Interventions: Dietary Supplement: Group 1 - diet rich in n-3 and n-6 PUFA
- Group 2 - diet rich in MUFA (Experimental): Assigned intervention: The dietary intervention was conducted by 60 days. Were prescribed normocaloric diets with similar macronutrient composition, varying only the type of lipids offered.
  Group 2 received diet rich in monounsaturated fatty acids (MUFA). The volunteers were asked to consume daily virgin olive oil, totaling 35.2g to 50.6g, and 1 capsule of 1g of soybean oil.
  Interventions: Dietary Supplement: Group 2 - diet rich in MUFA
- Group 3 - Placebo group (Experimental): Placebo group was instructed to keep their eating habits and consuming 1 sachet of 2g of soybean oil and 1 capsule of 1g of soybean oil by day.
  Interventions: Dietary Supplement: Group 3 - Placebo group

INTERVENTIONS:
Dietary Supplement: Group 1 - diet rich in n-3 and n-6 PUFA — In order to achieve the desired intake of unsaturated FA, the group received individual portions of vegetable oils in the form of sachets, which were consumed for lunch and dinner, besides gelatin capsules, for 60 days.
  Arms: Group 1 - diet rich in n-3 and n-6 PUFA
Dietary Supplement: Group 2 - diet rich in MUFA — In order to achieve the desired intake of unsaturated FA, the group received individual portions of vegetable oils in the form of sachets, which were consumed for lunch and dinner, besides gelatin capsules, for 60 days.
  Arms: Group 2 - diet rich in MUFA
Dietary Supplement: Group 3 - Placebo group — Placebo group was instructed to keep their eating habits and consuming placebo for 60 days.
  Arms: Group 3 - Placebo group

SUMMARY:
The purpose of this study is to determine whether the modulation of dietary lipids are effective in the treatment of obesity and comorbidities.

DETAILED DESCRIPTION:
Obesity is a complex disease of multifactorial etiology and difficult to control. Among lifestyle changes proposed to the treatment of this disease and comorbidities, there is the modulation of dietary lipid composition. This study aimed to evaluate the effects of the modulation of fatty acid (FA) polyunsaturated (PUFA) and monounsaturated (MUFA) in energy expenditure (EE), weight loss, body composition, lipid and glycemic profile, free fatty acids (FFA), glycerol, adiponectin, leptin, blood pressure (BP), feeding behavior and expression of PPARα and PPARγ2 genes in adipose tissue (AT) of obese women. It was conducted a parallel, randomized, controlled, single-blind study with dietary intervention (DI) for 60 days, where 32 women with obesity classes I and II were distributed into three groups: G1 = diet rich in n-3 PUFA and n-6 (n = 10); G2 = MUFA-rich diet (n = 11); and G3 = control (n = 11). For G1 and G2 were prescribed normocaloric diets with similar macronutrient composition, varying only the type of lipids offered. In order to achieve the desired intake of unsaturated FA, both groups received individual portions of vegetable oils in the form of sachets, which were consumed for lunch and dinner (G1 = mix of virgin olive oil [VOO] and soybean oil [SO], overall of 35.2g to 52.8g / day; G2 = VOO, overall of 35.2g to 50.6 g / day), besides gelatin capsules (G1 = 2 g of fish oil / day; G2 = 1 capsule of 1g of SO / day). G3 was instructed to keep their eating habits and consuming placebos (1 sachet of 2g of SO and 1 capsule of 1g of SO / day).

ELIGIBILITY:
Inclusion Criteria:

* obesity grades I and II (body mass index between 30 and 39,99 kg/m2);
* completion of basic education (former 4th primary series).

Exclusion Criteria:

* menopausal;
* weight loss more than three kilograms (3 kg) in the last three months;
* diagnosis of diabetes mellitus, heart disease, hypertension, nephropathy, liver diseases , thyroid dysfunction; gastrointestinal disorders , acquired immunodeficiency syndrome or cancer;
* cholecystectomy in the past 12 months and other recent surgeries;
* pregnancy or lactation;
* smokers;
* drugs to lipid-lowering, diabetes, hypertension, depression, or obesity;
* food history of allergy or intolerance to vegetable oils (olive oil, soy or canola), fish oil, fish and / or seafood.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Compare the effects of modulation of PUFA and MUFA in energy expenditure of obese women | Change from baseline energy expenditure at 2 months
  The energy expenditure was evaluated by indirect calorimetry (Vmax Encore 29 Systems®)

SECONDARY OUTCOMES:
Effects of modulation of PUFA and MUFA in body weight of obese women | Change from baseline loss of body weight at 2 months
Effects of modulation of PUFA and MUFA in body composition of obese women | Change from baseline body composition at 2 months
  The body composition was evaluated by electrical bioimpedance
Effects of modulation of PUFA and MUFA in feeding behavior of obese women | Change from baseline feeding behavior at 2 months
  Feeding behavior was evaluated by Three Factor Eating Questionnaire
Effects of modulation of PUFA and MUFA in gene expression of obese women | Change from baseline gene expression at 2 months
  Gene expression of PPARα and PPARγ2 in adipose tissue
Effects of modulation of PUFA and MUFA in blood glucose of obese women | Change from baseline blood glucose at 2 months
Effects of modulation of PUFA and MUFA in blood insulin of obese women | Change from baseline blood insulin at 2 months
Effects of modulation of PUFA and MUFA in insulin resistance of obese women | Change from baseline insulin resistance at 2 months
  Insulin resistance was evaluated by Homeostasis Model Assessment
Effects of modulation of PUFA and MUFA in insulin sensitivity of obese women | Change from baseline insulin sensitivity at 2 months
  Insulin resistance was evaluated by Quantitative Insulin Sensitivity Check Index
Effects of modulation of PUFA and MUFA in total cholesterol and fractions of obese women | Change from baseline total cholesterol and fractions at 2 months
  total cholesterol and fractions and triglycerides
Effects of modulation of PUFA and MUFA in adiponectin of obese women | Change from baseline adiponectin at 2 months
  serum adiponectin
Effects of modulation of PUFA and MUFA in leptin of obese women | Change from baseline leptin at 2 months
  serum leptin
Effects of modulation of PUFA and MUFA in TNF alpha of obese women | Change from baseline TNF alpha at 2 months
  serum TNF alpha
Effects of modulation of PUFA and MUFA in interleukin 6 of obese women | Change from baseline interleukin 6 at 2 months
  serum interleukin 6

CONTACTS AND LOCATIONS:
Overall Officials: Eliane L Rosado, Doctor, Study Director — UFRJ

REFERENCES:
- [Background] Ailhaud G, Massiera F, Weill P, Legrand P, Alessandri JM, Guesnet P. Temporal changes in dietary fats: role of n-6 polyunsaturated fatty acids in excessive adipose tissue development and relationship to obesity. Prog Lipid Res. 2006 May;45(3):203-36. doi: 10.1016/j.plipres.2006.01.003. Epub 2006 Feb 10. PMID 16516300
- [Background] Barson JR, Karatayev O, Gaysinskaya V, Chang GQ, Leibowitz SF. Effect of dietary fatty acid composition on food intake, triglycerides, and hypothalamic peptides. Regul Pept. 2012 Jan 10;173(1-3):13-20. doi: 10.1016/j.regpep.2011.08.012. Epub 2011 Sep 6. PMID 21903140
- [Background] Bjermo H, Iggman D, Kullberg J, Dahlman I, Johansson L, Persson L, Berglund J, Pulkki K, Basu S, Uusitupa M, Rudling M, Arner P, Cederholm T, Ahlstrom H, Riserus U. Effects of n-6 PUFAs compared with SFAs on liver fat, lipoproteins, and inflammation in abdominal obesity: a randomized controlled trial. Am J Clin Nutr. 2012 May;95(5):1003-12. doi: 10.3945/ajcn.111.030114. Epub 2012 Apr 4. PMID 22492369
- [Background] Buckley JD, Howe PR. Anti-obesity effects of long-chain omega-3 polyunsaturated fatty acids. Obes Rev. 2009 Nov;10(6):648-59. doi: 10.1111/j.1467-789X.2009.00584.x. Epub 2009 May 12. PMID 19460115
- [Background] Casas-Agustench P, Lopez-Uriarte P, Bullo M, Ros E, Gomez-Flores A, Salas-Salvado J. Acute effects of three high-fat meals with different fat saturations on energy expenditure, substrate oxidation and satiety. Clin Nutr. 2009 Feb;28(1):39-45. doi: 10.1016/j.clnu.2008.10.008. Epub 2008 Nov 17. PMID 19010571
- [Background] Clarke SD, Gasperikova D, Nelson C, Lapillonne A, Heird WC. Fatty acid regulation of gene expression: a genomic explanation for the benefits of the mediterranean diet. Ann N Y Acad Sci. 2002 Jun;967:283-98. PMID 12079856
- [Background] Clevenger HC, Stevenson JL, Cooper JA. Metabolic responses to dietary fatty acids in obese women. Physiol Behav. 2015 Feb;139:73-9. doi: 10.1016/j.physbeh.2014.11.022. Epub 2014 Nov 13. PMID 25446217
- [Background] DeFina LF, Marcoux LG, Devers SM, Cleaver JP, Willis BL. Effects of omega-3 supplementation in combination with diet and exercise on weight loss and body composition. Am J Clin Nutr. 2011 Feb;93(2):455-62. doi: 10.3945/ajcn.110.002741. Epub 2010 Dec 15. PMID 21159785
- [Background] Flint A, Helt B, Raben A, Toubro S, Astrup A. Effects of different dietary fat types on postprandial appetite and energy expenditure. Obes Res. 2003 Dec;11(12):1449-55. doi: 10.1038/oby.2003.194. PMID 14694208
- [Background] Guri AJ, Hontecillas R, Bassaganya-Riera J. Dietary modulators of peroxisome proliferator-activated receptors: implications for the prevention and treatment of metabolic syndrome. J Nutrigenet Nutrigenomics. 2008;1(3):126-35. doi: 10.1159/000112460. Epub 2008 Feb 20. PMID 19776622
- [Background] Krebs JD, Browning LM, McLean NK, Rothwell JL, Mishra GD, Moore CS, Jebb SA. Additive benefits of long-chain n-3 polyunsaturated fatty acids and weight-loss in the management of cardiovascular disease risk in overweight hyperinsulinaemic women. Int J Obes (Lond). 2006 Oct;30(10):1535-44. doi: 10.1038/sj.ijo.0803309. Epub 2006 Mar 21. PMID 16552404
- [Background] Krishnan S, Cooper JA. Effect of dietary fatty acid composition on substrate utilization and body weight maintenance in humans. Eur J Nutr. 2014 Apr;53(3):691-710. doi: 10.1007/s00394-013-0638-z. Epub 2013 Dec 22. PMID 24363161
- [Background] Liao FH, Liou TH, Shieh MJ, Chien YW. Effects of different ratios of monounsaturated and polyunsaturated fatty acids to saturated fatty acids on regulating body fat deposition in hamsters. Nutrition. 2010 Jul-Aug;26(7-8):811-7. doi: 10.1016/j.nut.2009.09.009. Epub 2009 Dec 22. PMID 20022469
- [Background] Nakamura MT, Yudell BE, Loor JJ. Regulation of energy metabolism by long-chain fatty acids. Prog Lipid Res. 2014 Jan;53:124-44. doi: 10.1016/j.plipres.2013.12.001. Epub 2013 Dec 18. PMID 24362249
- [Background] Mejia-Barradas CM, Del-Rio-Navarro BE, Dominguez-Lopez A, Campos-Rodriguez R, Martinez-Godinez Md, Rojas-Hernandez S, Lara-Padilla E, Abarca-Rojano E, Miliar-Garcia A. The consumption of n-3 polyunsaturated fatty acids differentially modulates gene expression of peroxisome proliferator-activated receptor alpha and gamma and hypoxia-inducible factor 1 alpha in subcutaneous adipose tissue of obese adolescents. Endocrine. 2014 Feb;45(1):98-105. doi: 10.1007/s12020-013-9941-y. Epub 2013 Apr 2. PMID 23546614
- [Background] van Dijk SJ, Feskens EJ, Bos MB, Hoelen DW, Heijligenberg R, Bromhaar MG, de Groot LC, de Vries JH, Muller M, Afman LA. A saturated fatty acid-rich diet induces an obesity-linked proinflammatory gene expression profile in adipose tissue of subjects at risk of metabolic syndrome. Am J Clin Nutr. 2009 Dec;90(6):1656-64. doi: 10.3945/ajcn.2009.27792. Epub 2009 Oct 14. PMID 19828712
- [Derived] Lopes MCODS, Kaippert VC, Crovesy L, de Carvalho DP, Rosado EL. Monounsaturated fat-rich diet reduces body adiposity in women with obesity, but does not influence energy expenditure and substrate oxidation: a parallel randomized controlled clinical trial. Eur J Clin Nutr. 2024 Apr;78(4):335-343. doi: 10.1038/s41430-024-01401-3. Epub 2024 Jan 12. PMID 38216647